CLINICAL TRIAL: NCT04643470
Title: A Phase 2, Multicenter, Randomized, Double Blind, Placebo Controlled Study to Evaluate the Safety and Efficacy of Zanubrutinib in Patients With Active Proliferative Lupus Nephritis
Brief Title: Zanubrutinib in Participants With Active Proliferative Lupus Nephritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BGB-3111-217; CTR20202662 (Other: ChinaDrugTrials)
Record Dates: First submitted 2020-11-18; First posted 2020-11-25 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Lupus Nephritis
MeSH Terms: conditions — Lupus Nephritis | interventions — zanubrutinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Zanubrutinib Low Dose (Experimental): Participants will receive zanubrutinib 40 mg twice daily (BID) for 72 weeks
  Interventions: Drug: Zanubrutinib
- Zanubrutinib High Dose (Experimental): Participants will receive zanubrutinib 160 mg twice daily (BID) for 72 weeks
  Interventions: Drug: Zanubrutinib
- Zanubrutinib Medium Dose (Experimental): Participants will receive zanubrutinib 160 mg once daily (QD) for 72 weeks
  Interventions: Drug: Zanubrutinib
- Placebo (Experimental): Participants will receive placebo to match zanubrutinib for 72 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Zanubrutinib — Administered as specified in the treatment arm
  Other Names: BGB-3111; Brukinsa
  Arms: Zanubrutinib High Dose; Zanubrutinib Low Dose; Zanubrutinib Medium Dose
Drug: Placebo — Placebo to match zanubrutinib
  Arms: Placebo

SUMMARY:
The primary objective of this study is to evaluate the efficacy of zanubrutinib added to standard of care as measured by complete renal response for participants with active proliferative lupus nephritis

ELIGIBILITY:
Key Inclusion Criteria:

1. Clinical diagnosis of SLE according to the Systemic Lupus International Collaborating Clinics 2012 criteria.
2. ISN/RPS 2003 Class III/IV lupus nephritis [Type III(A), III (A+C), IV (A), and IV (A+C)], with or without Class V, as confirmed by a renal biopsy.
3. Positive antinuclear antibodies, positive anti-dsDNA autoantibody, and/or positive anti Smith autoantibody at screening
4. Has 24-hour urine protein excretion > 1.0 g at screening.

Key Exclusion Criteria:

Exclusion criteria related to systemic lupus erythematous and other diseases:

1. Glomerulonephritis caused by reasons other than systemic lupus erythematous.
2. Sclerosis in >50% of glomeruli on renal biopsy.
3. Any other inflammatory diseases that might confound the assessments of efficacy, including but not limited to rheumatoid arthritis, myositis, vasculitis, or overlapping syndrome.
4. Severe extrarenal SLE, including but not limited to severe pulmonary arterial hypertension, severe myocarditis, severe central nervous system lupus (such as neuropsychiatric SLE, seizures, psychosis, transverse myelitis, central nervous system vasculitis and optic neuritis), etc.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 177 (Actual)
Dates: Start 2020-12-22 (Actual); Primary Completion 2024-02-26 (Actual); Study Completion 2024-08-26 (Actual)

PRIMARY OUTCOMES:
Proportion of participants with complete renal response | Week 49 Day 1

SECONDARY OUTCOMES:
Proportion of participants achieving complete renal response | Up to Week 73 Day 1
Proportion of participants achieving partial renal response | Up to Week 73 Day 1
Proportion of participants achieving overall renal response | Up to Week 73 Day 1
Time to first complete renal response | Up to Week 73 Day 1
  The time from the date of randomization to the date of the first complete renal response
Time to first overall renal response | Up to Week 73 Day 1
  The time from the date of randomization to the date of the first overall renal response
Change in total Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) score | Baseline to Week 49 Day 1
  SLEDAI-2K score is a systemic lupus erythematosus (SLE) activity index based on the presence of 24 features in 9 organ systems which ranges from 0 - 105, with higher scores indicating more severe features in participants in the past 30 days
Area under plasma concentration time curve (AUC) of zanubrutinib | Week 1 Day 1 and Week 5 Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Zhen Yao, MD, Study Director — BeiGene
Locations (44):
- China (44):
  - Anhui Provincial Hospital, Hefei, Anhui
  - Peking University Peoples Hospital, Beijing, Beijing Municipality
  - Peking University International Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Zhongshan Hospital Xiamen University, Xiamen, Fujian
  - Sun Yat Sen Memorial Hospital, Sun Yat Sen University (North), Guangzhou, Guangdong
  - Guangdong Provincial Peoples Hospital, Guangzhou, Guangdong
  - The First Affiliated Hospital, Sun Yat Sen University, Guangzhou, Guangdong
  - The Third Affiliated Hospital, Sun Yat Sen University, Guangzhou, Guangdong
  - Guangdong Province Traditional Chinese Medical Hospitsal, Guangzhou, Guangdong
  - Jiangmen Central Hospital, Jiangmen, Guangdong
  - Peking University Shenzhen Hospital, Shenzhen, Guangdong
  - The Second Peoples Hospital of Shenzhen, Shenzhen, Guangdong
  - Liuzhou Workers Hospital, Liuchow, Guangxi
  - The Peoples Hospital of Guangxi Zhuang Autonomous Region, Nanning, Guangxi
  - Guizhou Provincial Peoples Hospital, Guiyang, Guizhou
  - Hainan General Hospital, Haikou, Hainan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Renmin Hospital of Wuhan University, Wuhan, Hubei
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - General Hospital of Eastern Theater Command, Nanjing, Jiangsu
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Wuxi Peoples Hospital, Wuxi, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - The First Affiliated Hospital of Nanchang University Branch Donghu, Nanchang, Jiangxi
  - The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The Second Hospital of Jilin University, Changchun, Jilin
  - First Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - General Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - The Second Affiliated Hospital of Xian Jiaotong University, Xi'an, Shaanxi
  - The First Affiliated Hospital of Xian Jiaotong University, Xi'an, Shaanxi
  - Shandong Provincial Hospital, Jinan, Shandong
  - The Affiliated Hospital of Qingdao University Branch South, Qingdao, Shandong
  - Huashan Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality
  - Shanghai General Hospital, Shanghai, Shanghai Municipality
  - Second Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Sichuan Academy of Medical Sciences and Sichuan Provincial Peoples Hospital, Chengdu, Sichuan
  - The Second Affiliated Hospital of Tianjin Medical University, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Ningbo First Hospital, Ningbo, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes